CLINICAL TRIAL: NCT02732184
Title: A Phase 2 Dose-Escalation Study of AEB1102 (Co-ArgI-PEG) in Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome Refractory to Hypomethylating Agents
Brief Title: A Multiple Dose, Dose Escalation Trial of AEB1102 in Patients With AML or MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-100C
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- AEB1102 (Co-ArgI-PEG) administered via IV weekly. (Experimental): Co-ArgI-PEG modified human arginase I
  Interventions: Drug: Co-ArgI-PEG modified human arginase I

INTERVENTIONS:
Drug: Co-ArgI-PEG modified human arginase I
  Other Names: AEB1102

SUMMARY:
This is the first study of the safety of increasing dose levels of AEB1102 in patients with Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome. The study will also evaluate the amounts of AEB1102 in blood, the effects of AEB1102 on blood amino acid levels and the antitumor effects of AEB1102.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age 18 and older
* Diagnosis of AML or MDS according to the WHO criteria
* AML relapsed or refractory to at least one attempt at induction or subjects not candidates for aggressive induction regimens
* MDS refractory to treatment with HMA therapy or with recurrence or progression of MDS following a response to an HMA
* Has adequate organ function: AST and ALT < 3X the ULN, serum bilirubin < 2X the ULN, serum creatinine of < 2 mg/dL, or a calculated creatinine clearance of > 50 mL/minute
* ECOG Performance Score of 0 -2
* Recovered from the effects of any prior systemic therapy, radiotherapy or surgery
* Willing to use physician approved birth control method

Exclusion Criteria:

* Current CNS Leukemia
* Acute promyelocytic leukemia or AML with a t(15;17) (q22;q12) cytogenetic abnormality or Bcr/Abl positive leukemia
* < 60 days from ASCT; has chronic graft-versus host disease (GVHD) or requires continued treatment with systemic immunosuppressive agents
* Uncontrolled infection
* Known HIV, hepatitis B or hepatitis C.
* Other active malignancy that requires therapy
* If female, is lactating or breast feeding
* Hypersensitivity to PEG or other component of AEB1102 (Co-ArgI-PEG)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Recommended Phase 2 Dose | 4 weeks
  The dose level at which no more than 1/6 patients experiences dose-limiting toxicity

SECONDARY OUTCOMES:
Safety profile (changes in physical exam, laboratory measures, reported adverse events) | 4 Weeks
  changes in physical exam, laboratory measures, reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Aeglea BioTherapeutics, Inc.
Locations (10):
- United States (7):
  - Comprehensive Cancer Center at University of Michigan, Ann Arbor, Michigan
  - Washington University Medical School, St Louis, Missouri
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor Scott & White, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec